CLINICAL TRIAL: NCT04722055
Title: A Multicenter Clinical Trial of Human Multigene Methylation Detection Kit (Fluorescent PCR)
Brief Title: A Multicenter Clinical Trial of Stool-based DNA Testing for Early Detection of Colon Cancer in China
Status: Completed | Type: Observational
Sponsor: Creative Biosciences (Guangzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KLM2020-02
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2011-11

CONDITIONS: Colorectal Cancer; Advanced Adenocarcinoma; Hyperplastic Polyp; Colorectal Neoplasms; Digestive System Neoplasm; Neoplasms
Keywords: Colorectal Cancer; Colon Cancer; Stool DNA test; fecal DNA test; Methylation Biomarkers; Colonoscopy; Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Neoplasms; Neoplasms; Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples With DNA — Isolated human DNA from stool samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Single arm of continuously enrolled participants. All eligible participants will be included in the study according to the inclusion criteria. In addition to giving stool samples for multigene methylation test, eligible participants need to undergo colonoscopy examination and have their biopsies taken when necessary (gold standard).
  Interventions: Diagnostic Test: Multigene Methylation Detection Kit

INTERVENTIONS:
Diagnostic Test: Multigene Methylation Detection Kit — Eligible participants are required to take stool samples for multigene methylation detection and gene sequencing, undergo colonoscopy examination, and have a biopsy when necessary (gold standard).
  Other Names: Colosafe 2.0

SUMMARY:
According to data from Global Cancer Statistics 2018, colorectal cancer (CRC) ranks second in incidence and fifth in mortality among all cancers in China. The underlying neoplastic progression from adenoma to CRC endures up to 10 years, providing an extended window for CRC detection and screening. Currently, fecal occult blood test (FOBT) and colonoscopy are the main diagnostic and screening methods for CRC in Chinese clinical practice. However, due to low patients' compliance with colonoscopy and poor sensitivity of FOBT, a large proportion of CRC could not be effectively diagnosed and treated at early stage. Therefore, noninvasive fecal DNA detection approach with enhanced performance is urgently needed in clinic.

The aim of this trial is to evaluate effectiveness of the Human Multigene Methylation Detection Kit (Fluorescent PCR) for auxiliary diagnosis of colorectal cancer. By assessing the level of DNA methylation of certain genes in human stool, the test can indicate whether cancerous and precancerous lesions exist in the areas of colon and rectum.

DETAILED DESCRIPTION:
The multicenter clinical trial will be conducted using a single-blind method. Stool samples provided by participants will be evaluated by Human Multigene Methylation Detection Kit (Fluorescent PCR). The kit will be used to qualitatively detect methylation levels of multiple genes in human stool samples in vitro by using Quantitative Methylation Specific PCR (qMSP). The principle of the method is as follows. First, the target DNA in human stool is extracted by magnetic bead-capture technology and then treated with sodium bisulfite. The sequence of unmethylated DNA will be changed while that of the methylated DNA remains the same after sodium bisulfite treatment. Subsequently, qMSP is employed to detect methylation levels of target genes in addition to ACTB gene (a reference gene). Controls of ACTB gene with and without methylation are tested simultaneously. Result of qMSP is dichotomized as positive and negative based on Ct value obtained. The test result is then verified by Sanger sequencing and compared with that from colonoscopy examination and pathology report. The main evaluation indexes for test performance are sensitivity, specificity, consistency rate, kappa coefficient.

ELIGIBILITY:
Inclusion Criteria:

* Participants must also meet the following three criteria to be included in this study:

  1. To be 40 to 79 years old, regardless of gender;
  2. To participate voluntarily and sign Informed Consent Form;
  3. To satisfy any of the following three conditions:

     1. Patients with colorectal cancer confirmed or suspected by colonoscopy or pathological biopsy;
     2. Patients with gastrointestinal disease or normal population to be examined by colonoscopy;
     3. Patients who are planning to undergo colonoscopy or have colonoscopy results from other interfering diseases.

Exclusion Criteria:

* Patients with any of the following conditions shall be excluded:

  1. To have had radical resection of colorectal cancer before enrollment in this study;
  2. To have been deemed ineligible to participate in the study by the principal investigator due to various other reasons.

Ages: 40 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants aged 40-79 years old, regardless of gender or region, and those who meet the inclusion criteria for this clinical trial, are eligible to enroll at the designated clinical sites. Up to 1113 participants will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1273 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2022-01-19 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Sensitivity | Two years
  Sensitivity is the true positive fraction of participants with colorectal cancer.
Specificity | Two years
  Specificity is the true negative fraction of participants without colorectal cancer.
Consistency rate | Two years
  Consistency rate is the fraction of both true positive and negative diagnostic test results among all participants.
Kappa coefficient | Two years
  Kappa coefficient is the consistency analysis of the extent of agreement between the test results of Colosafe 2.0 and reference colonoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Xianrang Song, PhD, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No
We are carefully considering all applicable regulations and laws governing sharing of patients' data from China online with the global public.